CLINICAL TRIAL: NCT06631898
Title: Evaluation of Dermatological Safety of Test Products by 24 Hours Patch Test Under Complete Occlusion or Semi Occlusion or Open Patch on Adult Healthy Human Subjects.
Brief Title: To Check Dermatological Safety of Test Products by 24 Hours Patch Test on Adult Healthy Human Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Blossom Microbiotics LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NB240048-BM
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Normal Skin

STUDY DESIGN:
Intervention Model Description: Primary Irritation Patch Test Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SaaTwae Bio-Natural Moisturizing Cream (Experimental): A 0.04 gm of test products along with controls (negative and positive) will be applied on the back of subjects i.e. between the scapula and waist through Finn chamber patch.
  Interventions: Other: SaaTwae Bio-Natural Moisturizing Cream

INTERVENTIONS:
Other: SaaTwae Bio-Natural Moisturizing Cream — A 0.04 gm of test products along with controls (negative and positive) will be applied on the back of subjects i.e. between the scapula and waist through Finn chamber patch.

SUMMARY:
This is single-center, evaluator blinded study in healthy human subjects. single 24-hour application of sponsors provided test product along with positive and negative control will be kept in contact with the skin if subject under icclllusion or semi occlusion or open patch for at least 24 hours (± 2 hours). safety will be assed through the study by monitoring of adverse event A sufficient number 26 subject will be enrolled to get 24 completed the study. There are total three visits in this study and are optional visit pre-screening visit : Lactic Acid Stinging test& Modified Dr baumenn's skin type questionnaire. Visit 01: Screening, Enrollment, and Patch Application (Day 01) Visit 02: Patch Removal After 24 hours of Application & 30 ± 5 min irritation scoring upon patch removal Visit 03: 24 (± 2 hour) irritation scoring (Day 03) visit 04: subject will be contacted telephonically on Day 08 for any signs of irritation at patch application site. Follow-up visit for reactions if any to confirm recovery (optional deemed necessary) Irritation scoring at 168 ± 2 hours post-patch removal (Day 09)

ELIGIBILITY:
Inclusion Criteria:

* 1) Age: 18-65 years (both inclusive) at the time of consent. 2) Sex: Males and non-pregnant/non-lactating females (preferably equal number of males and females).

  3) Subject with normal Fitzpatrick skin type III to V (Human skin colour determination scale).

  4) Females of childbearing potential must have a self-reported negative pregnancy test.

  5) Subject who do not have any previous history of adverse skin conditions and are not under any medication likely to interfere with the results.

  6) Subject is in good general health as determined by the Investigator on the basis of medical history.

  7) Subjects is willing to maintain the test patches in designated positions for 24 Hours.

  8) Subject is willing and able to follow the study directions, to participate in the study, returning for all specified visits.

  9) Subject must be able to understand and provide written informed consent to participate in the study.

  10) Subject is willing to refrain from vigorous physical exercise during the study period and follow all the instruction given.

Exclusion Criteria:

* 1) Subject having skin irritation, blemishes, excessive hair, moles, pigmentation, pimples, marks (e.g. tattoos (within the previous 3 months), scars, sunburn), open wounds, cuts, abrasions, irritation symptoms or any dermatological condition on the test site(s) i.e. back that can interfere with the reading.

  2) Medication which may affect skin response and/or past medical history. 3) Subject having history of diabetes 4) Subject have history of mastectomy for cancer involving removal of lymph nodes within the past year, or treatment of any type of cancer within the last 6 months.

  5) Subject suffering from any active clinically significant skin diseases which may contraindicate.

  6) Subject having history of any skin diseases including eczema, atopic dermatitis or active cancer.

  7) Participation in any patch test for irritation or sensitization within the last four weeks.

  8) Subject having history of asthma or COPD (Chronic obstructive pulmonary disease).

  9) Use of any: i. Prescribed or over-the-counter (OTC) anti-inflammatory drug within five (5) days prior to application.

ii. Antihistamine medication or immunosuppressive drugs within seven (7) days prior to first patch application.

iii. Systemic or topical corticosteroids at patch site within four (4) weeks of test product application (steroidal nose drops and/or eye drops are permitted) 10) Topical drugs used at application site. 11) Subject with Self-reported Immunological disorders such as HIV positive, AIDS and/or systemic lupus erythematous.

12) Individual who has a medical condition or is taking or has taken a medication which, in the Investigator's judgment, makes the subject ineligible or places the subject at undue risk.

13) Subject with known allergy or sensitization to medical adhesives, bandages. 14) Participation in other patch study simultaneously.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the dermatological safety of the test products by 24 Hours Patch Test | Irritation Scoring at T30 minutes and 24 hours post patch removal. Scoring can be done at T168 hours post-patch removal if needed.
  Dermatological safety of the test products by 24 Hours Patch Test will be evaluated by 0: No reaction and 4 Severe Reaction

SECONDARY OUTCOMES:
Safety of the skin | At T30 minutes and 24 hours post patch removal. Scoring can be done at T168 hours post-patch removal if required.
  To evaluate the Safety of the skin by visual dermatological assessment by 0: No reaction and 4 Severe Reaction

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, Principal Investigator — NovoBliss Research Pvt Ltd
Locations (1):
- NovoBliss Research Pvt.Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No